CLINICAL TRIAL: NCT02559843
Title: Effects of Pomegranate Juice Consumption on Glycemic Control, Lipid Profile, Oxidative Stress and Blood Pressure in Patients With Type 2 Diabetes
Brief Title: Effects of Pomegranate Juice on Oxidative Stress in Patients With type2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Faculty member, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 611
Record Dates: First submitted 2015-09-15; First posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes Type 2
Keywords: pomegranate; diabetes; oxidative stress
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pomegranate juice (Experimental): 200 ml pomegranate juice + lifestyle modification
  Interventions: Dietary Supplement: pomegranate juice
- control (Active Comparator): lifestyle modification including dietary recommendations
  Interventions: Behavioral: lifestyle modification

INTERVENTIONS:
Dietary Supplement: pomegranate juice
  Arms: pomegranate juice
Behavioral: lifestyle modification
  Arms: control

SUMMARY:
Introduction: Diabetes mellitus a chronic diseases, is the most common and important metabolic disease in human. Increased free radicals production due to hyperglycemia produces oxidative stress which worsens the disease and its complications. Pomegranate juice has antioxidant and antiatherosclerotic properties. The present study was planned to evaluate the effects of pomegranate juice consumption on glycemic control, lipid profile,blood pressure and oxidative stress in patients with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Age of 40-65 years
* Body Mass Index 18.5-30
* Fasting blood glucose ≥ 126 mg/dl

Exclusion Criteria:

* Smoking
* insulin for blood glucose control
* taking estrogen or progesterone (if female)
* Taking antioxidant supplements
* suffering from any other chronic diseases
* Participants are also excluded if they missed more than 10% of their pomegranate juice packs

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
total antioxidant capacity | 6 weeks

SECONDARY OUTCOMES:
fasting blood glucose | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- NNFTRI clinic, Tehran, Tehran Province, Iran